CLINICAL TRIAL: NCT04403061
Title: Th1/Th2/Th17/TREG Response and TLRs Activation/KIR Receptors for Predicting the Evolution of the SARS Cov-2 Infected Patients
Brief Title: Th1/Th2/Th17/TREG and TLRs Activation/KIR for COVID 19 Prediction of Outcome
Acronym: Resistir
Status: Completed | Type: Observational
Sponsor: Asociacion para el Estudio de las Enfermedades Infecciosas (Network)
Collaborators: Fundacion para la Investigacion Biomedica del Hospital Universitario Ramon y Cajal (Other)
Responsible Party: Sponsor
Other Study IDs: EC128/20
Record Dates: First submitted 2020-05-23; First posted 2020-05-27 (Actual); Last update posted 2021-01-12 (Actual); Status verified 2021-01

CONDITIONS: Disease, Viral; Cytokine Release Syndrome; TLRs
MeSH Terms: conditions — Virus Diseases; Cytokine Release Syndrome | interventions — Immunity, Cellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Cytokines measurement — Quantification of plasma cytokine levels of human GM-CSF, IFN-α, IFN-γ, IL-2, IL-4, IL-5, IL-6, IL-9, IL-10, IL-12p70, IL-17A, and TNF-α using multiplex technol-ogy (quantitative measure).
Diagnostic Test: Cellular response — SARS-CoV-2 peptides (Prot-S, Pros-N and Port-M) will be used to activate CD4 and CD8 T cells. Cytokines released, such as IFNg, TNFa, IL4, IL17A, and IL2, from each cell subset will be measured by flow cytometry (quantitative measure).
Diagnostic Test: TLRs activation measurement — After specific cell activation through TLR7/8 receptors, such as resiquimod, ORN R-0002, ORN R-0006, ORN R-1263, ORN R-2336, and controls as Poly (I:C), the release of IFNa, IFNg, TNFa, IL12, and IL6 will be analyzed (quantitative measure).
Diagnostic Test: KIR phenotype evaluation — Characterization of the presence of 14 genes plus 2 pseudogenes of KIR gene family (qualitative genotyping) by PCR, mRNA expression profiling (quantitative measures) by RT-PCR, and phenotyping of human NK cells analyzing different KIR receptors (quantitative measure) by flow cytometry, will be analyzed.

SUMMARY:
To ascertain globally the changes in the cytokines involved and TLRs/KIR activation in patients admitted to the hospital with a COVID-19 diagnosis, and the changes after initiation of the different therapies

DETAILED DESCRIPTION:
COVID-19 is a disease with an initial viral phase followed, usually at the 7th day, of an inflammatory state (cytokine storm) leading to respiratory distress, ICU admission and risk of death. Thus, several biological agents, antagonists of the different cytokines (IL-6, IL-1) have been used for patients with severe disease. However, there are no data about the cytokine changes, at admission and after therapy, and its predictive value, a fundamental knowledge to establish the best therapeutic strategy.

The first line of immune defense is the interaction of the virus with innate immunity cell members. The toll like receptors (TLRs) family is a group of pattern recognition receptors that include many different molecules (21-23). These bindings can activate dendritic cells, monocytes, macrophages. There is an important RNA and DNA connection, activation of TLRs, the production of type I interferons, and the development of some autoimmune diseases. TLR7 and TLR8 specifically recognize simple-chain RNA of viruses and are expressed in endosomal membranes. TLR8 is expressed in regulatory cells (Treg) and its activation results in inhibition of its regulatory functions. Natural killer cells (NK) respond to alterations of class I HLA molecules present in infected cells (24-26). An increase in class I HLA expression could lead to an increase in NK activation by increasing its ability to produce IFN-gamma. Therefore, the reasons for KIR binding are often variable between individuals and between populations.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of COVID-19 (PCR confirmed)

Exclusion Criteria:

* No informed consent
* Presence of chronic therapy with immunomodulators, corticoids or antineoplastic agents.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a diagnosis of COVID-19
Sampling Method: Non-Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2020-05-22 (Actual); Primary Completion 2020-12-22 (Actual); Study Completion 2021-01-10 (Actual)

PRIMARY OUTCOMES:
Changes in cytokines associated with SARS CoV-2 infection | 1 month
Evaluation of cellular response | 1 month
TLRs activation | 1 month
KIR phenotype determination | 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Ramon y Cajal, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided
Pending to establish collaboration to share cytokine measurements